CLINICAL TRIAL: NCT05418881
Title: Evaluation and Implementation of Mobile Tracking Devices to Increase Safety in Hospitalized Patients - MONITOR 2022
Brief Title: Evaluation and Implementation of Mobile Tracking Devices to Increase Safety in Hospitalized Patients (MONITOR)
Acronym: MONITOR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: University of Wuerzburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: MONITOR 2022
Record Dates: First submitted 2022-05-18; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Fitness Trackers; Hemodynamic Monitoring; Internet of Things; Postoperative Complications; Wearable Electronic Devices; Anesthesia; Surgery
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- postoperative Spot Measurements (Other): Measurement of vital signs via 4 different tracking devices in the setting of post-anaesthesia care unit. Simultaneous collection of vital signs measured by the gold standard of clinical monitoring (ecg, blood-gas-analysis, invasive blood pressure, transmissive photoplethysmography).
  Interventions: Device: Mobile Tracking Device (one spot)
- Longitudinal postoperative Measurements (Other): Continuous measurement of vital signs and activity level with tracking devices for the postoperative period in the patient ward up until 21 days postoperative.
  Interventions: Device: Mobile Tracking Device (one spot); Device: Mobile Tracking Device + Activity Sensor (longitudinal)

INTERVENTIONS:
Device: Mobile Tracking Device (one spot) — Patients will be fitted with 4 different tracking devices (Garmin Fenix 6 Pro®, Apple Watch 7®, FitBit Sense®, Withings ScanWatch®).
Device: Mobile Tracking Device + Activity Sensor (longitudinal) — Patients will be fitted with 1 of 3 different tracking devices (Garmin Fenix 6 Pro®, Apple Watch 7®, Withings ScanWatch®). The type of tracking device will be randomized. Additionally an Activity Tracker and one-channel ECG (Movesense®) will be worn by the patients.
  Arms: Longitudinal postoperative Measurements

SUMMARY:
The study investigates the technical feasibility of using mobile health trackers for monitoring of hospitalized patients. Therefore the measurement accuracy of several vital parameters in postoperative hospitalized patients will be compared to clinical gold standard. Factors that could have an influence on the measurement accuracy of the mobile sensors will be investigated.Furthermore patient compliance in continous use of mobile health trackers and technical feasibility of needed data flow will be analyzed. In addition, patients' activity levels are recorded and correlated with various clinical parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients with elective surgery (≥ 18 years).
* Written informed consent to participate in the study
* Planned invasive arterial blood pressure measurement

Exclusion Criteria:

* Postoperative invasive ventilation
* American Society of Anaesthesiologists (ASA) Class V
* Outpatient surgical procedure
* Previous participation in this study
* Patients unable to give consent or patients who do not have adequate German language skills
* Suspected lack of compliance
* Skin lesions of the forearms or inability to wear a tracking device
* Known allergy to latex/silicone/nickel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Measurement accuracy | postoperative until hospital discharge up to 21 days
  Heart rate as compared to ECG
Measurement accuracy | postoperative until hospital discharge up to 21 days
  Oxygen saturation as compared to arterial blood gas analysis

SECONDARY OUTCOMES:
Patient compliance with mobile tracking devices | postoperative until hospital discharge up to 21 days
  As measured by a survey
Postoperative inertial movement | postoperative until hospital discharge up to 21 days
  As measured by an inertial activity sensor (MoveSense®) in "inertial measurement units" (IMU)
Postoperative step count | postoperative until hospital discharge up to 21 days
  As measured by tracking devices in steps per day

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Meybohm, Prof. Dr., Study Director — Wuerzburg University Hospital
Locations (1):
- Wuerzburg University Hospital, Würzburg, Bavaria, Germany

REFERENCES:
- [Derived] Helmer P, Hottenrott S, Rodemers P, Leppich R, Helwich M, Pryss R, Kranke P, Meybohm P, Winkler BE, Sammeth M. Accuracy and Systematic Biases of Heart Rate Measurements by Consumer-Grade Fitness Trackers in Postoperative Patients: Prospective Clinical Trial. J Med Internet Res. 2022 Dec 30;24(12):e42359. doi: 10.2196/42359. PMID 36583938